CLINICAL TRIAL: NCT01646008
Title: Correlation Between Carbon Dioxide Measured in End of Exhalation and Arterial Blood in Chronic Obstructive Pulmonary Disease (COPD) in Intensive Care Unit With Nasal Cannula
Brief Title: Correlation Between Carbon Dioxide Measured in End of Exhalation and Arterial Blood
Status: Completed | Type: Observational
Sponsor: Hospital Universitario Getafe (Other)
Responsible Party: Principal Investigator, Susana Arias Rivera, Registered Nurse, Hospital Universitario Getafe
Other Study IDs: Carbon dioxide Getafe
Record Dates: First submitted 2012-07-18; First posted 2012-07-20 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Correlation Between Exhaled Carbon Dioxide and in Arterial Blood

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- respiratory
  Interventions: Other: To measure carbon dioxide by capnography and arterial blood

INTERVENTIONS:
Other: To measure carbon dioxide by capnography and arterial blood — Three times per day will be measured exhaled carbon dioxide and obtained in arterial blood sample.
Other: to measure carbon dioxide by capnography and arterial blood — three times per day we will obtained arterial blood samples and measurements of carbon dioxide by capnography

SUMMARY:
The purpose of this study is to study the correlation between carbon dioxide measured by capnography at the enf of exhalation and arterial blood in COPD patients with nasal cannula in critical care unit.

ELIGIBILITY:
Inclusion Criteria:

* Adults
* COPD patients

Exclusion Criteria:

* Under-aged
* Pregnant
* Major burns

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult COPD patients admitted to the ICU who consent
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2012-04; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susana Arias-Rivera, Graduate, Principal Investigator — Hospital Universitario de Getafe, Spain
Locations (1):
- Hospital Universitario de Getafe, Getafe, Madrid, Spain